CLINICAL TRIAL: NCT02637336
Title: Acute Cardiovascular Responses in Hypertensive Individuals
Brief Title: Study to Investigate Effects of Different Therapies for the Treatment of Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do vale do São Francisco (Other)
Collaborators: Fundação de Amparo à Ciência e Tecnologia de Pernambuco (Other)
Responsible Party: Principal Investigator, Marcus Amando Fernandes da Silva, Master's Degree student, Universidade Federal do vale do São Francisco
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UNIVASF
Record Dates: First submitted 2015-12-14; First posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Hypertension
Keywords: Therapies. Autonomic nervous system. Cardiovascular stress
MeSH Terms: conditions — Hypertension | interventions — Acupuncture Therapy; Aromatherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Acupuncture (Experimental): acupuncture session were inserted, and maintained for 20 minutes in paragraph 6 of the channel the pericardium (Neiguan).
  Interventions: Device: Acupuncture
- Aerobic Exercise (Experimental): The aerobic exercise session was conducted through 20 minutes.
  Interventions: Device: Aerobic exercise
- Aromatherapy (Experimental): Eucalyptus essential oil was inhaled by volunteers for 20 minutes
  Interventions: Device: Aromatherapy
- Control (No Intervention): In the control session the volunteers remained seated at rest for 20 minutes without performing therapy.

INTERVENTIONS:
Device: Acupuncture — Acupuncture in point 6 of the pericardium channel (neiguan) bilaterally
  Arms: Acupuncture
Device: Aerobic exercise — aerobic exercise of moderate intensity
  Arms: Aerobic Exercise
Device: Aromatherapy — inhalation of eucalyptus essential oil
  Arms: Aromatherapy

SUMMARY:
The aim of this study was to evaluate the acute cardiovascular responses in hypertensive individuals, in waking and sleeping periods after application of different non-pharmacological therapies for the control of blood pressure (BP). Randomly and random volunteers held a session of each therapy: Acupuncture, aerobic exercise, essential oil inhalation, and session control with a minimum interval of 72 hours between them. On the day of sessions the volunteers did not use antihypertensive medication. The variables measured in the survey were the blood pressure and heart rate variability (HRV). Descriptive statistical averaging procedures, standard deviation and standard error of mean were adopted. Two-way ANOVA for repeated measures was performed post-hoc Tukey. The level of the study significance was set at p <0.05.

DETAILED DESCRIPTION:
This study deals with a controlled trial and randomized crossover, with intentional non-probabilistic sample. All participants were informed of the procedures adopted in the research, and then signed the Informed Consent and Informed (IC) according to the resolution 466/12 of the National Health Council (Annex 1). The initial recruitment of volunteers was held in October 2014 with the initial assessments being carried out in the same month, after the project is approved by the Ethics Committee and Ethics Studies and Research of the Federal University of São Francisco Valley under the registration number 0010 / 240914 CEDEP / UNIVASF, and data collection with volunteers was completed in July 2015.

The plant material of Eucalyptus globulus was collected in January and May 2015 in the city Petrolina, Pernambuco state, Brazil. The process of extraction of essential oil of eucalyptus, made by hydrodistillation method by Clevenger system. To set the number of survey participants was conducted sample calculation by G.Power 3.0 program where the F test was chosen - two-way ANOVA for repeated measures between groups and within the group. Whereas four (04) experimental sessions and eighteen (18) measures time for each session, as well as α = 0.05 and power = 0.80, the sample size of 12 subjects was required.

Participants were randomly recruited in health centers in the city of Petrolina / PE through disclosure / meeting to present the research project, in addition to the collaboration of health workers from surrounding neighborhoods to UNIVASF.

All participants were divided into blocks in accordance with CONSORT criteria. Initially, the research project, along with the IC, was presented to each of the candidates to volunteer, with discussion of the risks and benefits, both scientific and individual would be likely to compose the study sample. After agreeing on participation, and application of history about health history, readiness for exercise and risk stratification according to guidelines from the American College of Sports Medicine, the informed consent was signed, and then scheduled with the volunteer the day and time of the completion of resting ECG examination (held in a large hospital in Petrolina / PE and funded by the researchers), to check for possible abnormalities and ischemia suggestion above or below unevenness in the ST segment> 2 mm or inversion of the T wave. All ECG's 12-lead were performed and evaluated by a cardiologist, where no examination apesentou suggestion ischemia or abnormality that would prevent volunteer to carry out all stages of safely search. After meeting and selection of the sample in accordance with the guidelines on inclusion profile, participants were invited to attend the morning to CEFIS of UNIVASF to carry out the anthropometric measurements (height, weight, body mass index, waist circumference and body fat percentage), and schedule for the start of the experimental sessions.

Volunteers had the orientation to suspend the anti-hypertensive medication on the day of each session, and only return to use after the removal of equipment (next day) by the researcher. In addition to this recommendation, the volunteers should not eat on the day of the interventions, substances that contain caffeine, alcohol, chocolate, tea, passion fruit or any other stimulant or CNS retardant, but the eating routine should be followed. The practice of physical activity, including sexual, was banned in the days that applied sessions.

On different days, with an interval of at least 72 hours, and in a randomized order, acupuncture, aerobic exercise, inhalation of essential oil of eucalyptus, and control were applied. In order to minimize the influence of the circadian rhythm, the sessions were always made at the same time of day (between 8 am and 9 am). Each treatment lasted for twenty (20) minutes. The living laboratory procedures was controlled temperature between 23 ° C and 24 ° C for all sessions.

The acupuncture session (ACUP) were placed, and maintained for 20 minutes so perpendicularly to the skin, two specific needles, stainless steel, sterilized and disposable (one on each arm) of 0.25mm brand Dongbang x 0.30 mm, in Section 6 of the pericardium channel (Neiguan), located 2 tsun (approximately 5 cm) proximal to the crease of the wrist, ventral aspect.

The aerobic exercise session (EXER) was conducted through 20-minute walk or jog on a treadmill of CEFISE brand, model TK30 (Campinas, BRA). The intensity was equivalent to 60% of the RHR (maximal HR - resting HR x 0.6 + HR rest).

In session eucalyptus essential oil (OIL) the subject sat, as in the rest time, and remained breathing naturally for 20 minutes with a disposable face mask, soaked in 0.25 ml of essential oil of eucalyptus measured by Adjustable Pipettor Kacil DSA ® Model 100 / 1000μl.

The session control (CONT) volunteers remained seated on standing for 20 minutes in the same manner and same chair used in acupuncture and inhalation of essential oils, but without performing any treatment.

The BP was assessed by ABPM device brand Meditech ABPM-04 (Micromed, BRA). The contents of the BP analyzed in this study were: systolic BP (SBP); Diastolic BP (DBP); BP Average (PAM), as follows: MAP = DAP + [(PAS-DAP) / 3]; Pressure overload (percentage> 125/75 mmHg in 24 hours;> 130 / 85mmHg in the Vigil and> 110/70 in Sleep, respectively for SBP and DBP); Night decline (relative percentage difference between the average sleep BP and the BP in the wake average). The measurements were taken every 15 minutes during daytime and every 30 minutes during sleep.

HRV was analyzed through the records of RRi intervals obtained by heart rate monitor brand Polar RS800CX model (Polar Electro Oy, FI-90440 KEMPELE, Finland) and this validated equipment and high reproducibility. The HRV indexes were analyzed by linear methods in the time domain (RRi, RMSSD, pNN50) and frequency (LF, HF and LF: HF), and the non-linear method by the standard deviation of RRI intervals (SD1). Records of RRi series were captured and recorded on the watch belonging to the equipment, continuously throughout the period of the day after the session, and analyzed using the software Kubios v. 2.0 at intervals of 5 minutes.

Descriptive statistical averaging procedures, standard deviation (SD) and standard error of the mean (SEM) was adopted. Shapiro-Wilk test for normality analysis was used, and in case of normality given a two-way ANOVA for repeated measures was performed post-hoc Tukey. For non-parametric data we used nonparametric ANOVA for analysis. The level of the study significance was set at p <0.05, using the Statistica software version 7.0.

ELIGIBILITY:
Inclusion Criteria:

* hypertensive mens;
* clinically stable.

Exclusion Criteria:

* Abnormalities in Resting ECG with cardiac ischemia suggestion;
* Rank in Category 3 (known serious illness) the risk stratification of the American College of Sports Medicine;
* Use of beta blocker medicine;
* Heart or kidney failure;
* Stroke history, coronary or peripheral arterial disease;
* Decompensated diabetes with blood glucose greater than 300 mg.dL-1;
* Autonomic dysfunction or severe peripheral;
* Any amputation of limbs; Regular physical activity practice (> 150 minutes per week) in the last 06 months;
* Uncontrolled hypertension with systolic blood pressure above 160 mmHg and diastolic blood pressure above 105 mmHg without medication;
* Abnormality in the blood coagulation;
* Allergy to the material of the acupuncture needle (stainless steel).

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Blood pressure outside the laboratory | 16 hours

SECONDARY OUTCOMES:
Blood pressure in the laboratory | 02 hours
Heart rate variability in the laboratory | 02 hours
Heart rate variability outside the laboratory | 16 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marcus AF Silva, Principal Investigator — UNIVASF